CLINICAL TRIAL: NCT00608998
Title: Vascular Risk Factors and Coronary Calcifications in Chronic Renal Failure Patients: Identification of Specific Factors Linked to Renal Failure Progression
Brief Title: Identification of Cardiovascular Risk Factors Linked to Renal Failure Progression
Acronym: Pre-HD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 7853
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2008-01

CONDITIONS: Chronic Renal Failure
Keywords: Chronic renal failure; Vasculopathy; Cardiovascular risk; Chronic renal failure patients
MeSH Terms: conditions — Kidney Failure, Chronic; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood white cells serum plasma urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to appreciate the influence of renal failure progression on vasculopathy (coronary calcifications and left ventricular hypertrophy) and cardiovascular risk factors.

DETAILED DESCRIPTION:
The aim of this study is to appreciate the relationship between:

* extension of coronary calcifications and chronic renal failure progression
* extension of coronary calcifications and levels of osteoprotegerin (bone disease marker)
* cardiovascular risk factors and coronary calcifications
* cardiovascular risk factors and existence of cardiovascular diseases

ELIGIBILITY:
Inclusion Criteria:

* Patient who has signed the written consent form
* Patient aged > 18 and < 90 years
* Chronic renal failure defined by glomerular filtration rate (GFR)

  * group 1: GFR >90 mL/min with urinary biological abnormalities and GFR comprised between 90 and 60 mL/min
  * group 2: GFR comprised between 60 and 30 mL/min
  * group 3: GFR <30 mL/min but without dialysis therapy

Exclusion Criteria:

* Chronic renal failure patient requiring dialysis therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
description of osteoprotegerin levels according to chronic renal failure progression | inclusion

SECONDARY OUTCOMES:
calcium score description according to chronic renal failure progression | inclusion
osteoprotegerin description according to calcium score | inclusion
relationship between cardiovascular risk factors and calcium score | inclusion
relationship between cardiovascular risk factors and cardiovascular disease | inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Bernard CANAUD, Pr, Principal Investigator — CHU Lapeyronie Montpellier France; Jean-Paul CRISTOL, Pr, Study Chair — CHU Lapeyronie Montpellier France; Hélène VERNHET, Pr, Study Chair — CHU Arnaud de Villeneuve Montpellier France; Kada KLOUCHE, Dr, Study Chair — CHU Lapeyronie Montpellier France; Hélène LERAY-MORAGUES, Dr, Study Chair — CHU Lapeyronie Montpellier France
Locations (1):
- Centre Hospitalier Universitaire, Montpellier, France